CLINICAL TRIAL: NCT00590694
Title: Determining Optimal Treatment Algorithms for Macular Degeneration Pigment Epithelial Detachments Treated With Intraocular Lucentis
Brief Title: Lucentis for Age-related Macular Degeneration Pigment Epithelial Detachments
Acronym: DETAIL
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pacific Eye Associates (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DETAIL Study for PED in AMD
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Last update posted 2012-04-12 (Estimated); Status verified 2012-04

CONDITIONS: Age-related Macular Degeneration; Pigment Epithelial Detachment; Neovascular Macular Degeneration; Wet Macular Degeneration
Keywords: ranibizumab; Lucentis; Pigment Epithelial Detachment; Macular Degeneration; PrONTO
MeSH Terms: conditions — Macular Degeneration; Retinal Detachment; Wet Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group1 (Active Comparator): Will receive ranibizumab treatments until resolution of macular edema only and as macular edema recurs.
  Interventions: Drug: ranibizumab
- Group 2 (Active Comparator): Will receive ranibizumab treatments until resolution of both macular edema and PED, and as macular edema or PED recur.
  Interventions: Drug: ranibizumab

INTERVENTIONS:
Drug: ranibizumab — 0.5mg injection monthly according to protocol for one year
  Other Names: Lucentis injection

SUMMARY:
Patients with neovascular Age-related macular degeneration (AMD) and the particular feature of pigment epithelial detachments (PEDs) were not studied in the Phase III trials for ranibizumab (Lucentis). The PrONTO study was the first ranibizumab study to enroll such patients but only treated with ranibizumab until fluid within the layers of the retina was absent, not until the entire PED was absent. This study hypothesizes that there may be a difference in benefit between patients treated until just the retinal edema is gone and those in which the retinal edema and PED are both gone.

ELIGIBILITY:
Inclusion Criteria:

* Neovascular age-related macular degeneration patients over age 50
* Presence of a pigment epithelial detachment on optical coherence tomography
* Initial or recurrent disease
* Previous treatment allowed
* Visual acuity between Snellen 20/40 - 20/400

Exclusion Criteria:

* More than three previous treatments with PDT or other radiation/laser therapy
* Previous vitrectomy or other AMD surgical intervention
* Severe scarring or severe concurrent ocular disease (uncontrolled glaucoma)

Patients eligible for the study are randomized into one of two groups. Group 1 receives injections of ranibizumab until retinal edema is resolved. Group 2 receives ranibizumab injections until both retinal edema and the PED are resolved. Study duration is one year with visits once per month.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Mean change in visual acuity from baseline over 12 months | 12 months

SECONDARY OUTCOMES:
Time to OCT resolution of macular edema and pigment epithelial detachment | One year
Proportion of patients with complete resolution of PED at 6 and 12 months | 12 months
Durability of outcome: time from last ranibizumab injection to retreatment | One year

CONTACTS AND LOCATIONS:
Overall Officials: Anne Fung, MD, Principal Investigator — Pacific Eye Associates / California Pacific Medical Center
Locations (1):
- Pacific Eye Associates, San Francisco, California, United States

REFERENCES:
- [Background] Fung AE, Lalwani GA, Rosenfeld PJ, Dubovy SR, Michels S, Feuer WJ, Puliafito CA, Davis JL, Flynn HW Jr, Esquiabro M. An optical coherence tomography-guided, variable dosing regimen with intravitreal ranibizumab (Lucentis) for neovascular age-related macular degeneration. Am J Ophthalmol. 2007 Apr;143(4):566-83. doi: 10.1016/j.ajo.2007.01.028. PMID 17386270
- See also: Pacific Eye Associates website — http://www.pacificeye.com/